CLINICAL TRIAL: NCT05002192
Title: A Retrospective, Real-world Study of Eucalyptol, Limonene and Pinene Enteric Soft Capsules Used in the Expectorant Treatment of Community-acquired Pneumonia
Brief Title: A Retrospective, Real-world Study of ELP Used in the Expectorant Treatment of Community-acquired Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Grand Johamu Pharmaceutical Company, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: YD_SMQD_ELP_202009
Record Dates: First submitted 2021-07-12; First posted 2021-08-12 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-07

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Eucalyptol; Limonene; Ambroxol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- ELP_ONLY: Patients who were diagnosed with community-acquired pneumonia and were treated with Eucalyptol, Limonene and Pinene Enteric Soft Capsules, not treated with other oral mucolytics.
  Interventions: Drug: Eucalyptol, Limonene and Pinene Enteric Soft Capsule
- EXP_ONLY: Patients diagnosed with community-acquired pneumonia and treated with an oral mucolytic drug other than Eucalyptol, Limonene and Pinene Enteric Soft Capsules.
  Interventions: Drug: Other oral mucolytic drugs
- ELP+AMB: Patients diagnosed with community-acquired pneumonia and treated with Eucalyptol, Limonene and Pinene Enteric Soft Capsules and ambroxol injection.
  Interventions: Drug: Eucalyptol, Limonene and Pinene Enteric Soft Capsule; Drug: Ambroxol injection
- EXP+AMB: Patients diagnosed with community-acquired pneumonia and treated with oral mucolytics and ambroxol injection other than Eucalyptol, Limonene and Pinene Enteric Soft Capsules.
  Interventions: Drug: Ambroxol injection; Drug: Other oral mucolytic drugs
- AMB_ONLY: Patients diagnosed with community-acquired pneumonia and treated with ambroxol injection alone.
  Interventions: Drug: Ambroxol injection

INTERVENTIONS:
Drug: Eucalyptol, Limonene and Pinene Enteric Soft Capsule — Compare the efficacy, safety and economic evaluation of pneumonia expectorant treatment in the cohort of ELP_ONLY and EXP_ONLY cohort
  Groups: ELP+AMB; ELP_ONLY
Drug: Ambroxol injection — Compare the efficacy, safety and economic evaluation of pneumonia expectorant treatment in the cohort of ELP+AMB and cohort EXP+AMB Compare the efficacy, safety and economic evaluation of pneumonia expectorant treatment in the cohort of ELP+AMB and AMB_ONLY cohort Compare the efficacy, safety and economic evaluation of pneumonia expectorant treatment in the cohort of ELP+AMB and AMB_ONLY cohort
  Groups: AMB_ONLY; ELP+AMB; EXP+AMB
Drug: Other oral mucolytic drugs — Compare the efficacy, safety and economic evaluation of pneumonia expectorant treatment in the cohort of ELP_ONLY and EXP_ONLY cohort
  Groups: EXP+AMB; EXP_ONLY

SUMMARY:
Through a series of retrospective analysis, it is hoped that an objective evaluation of the effect and safety of Eucalyptol, Limonene and Pinene Enteric Soft Capsules in the treatment of community-acquired pneumonia can be made.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with community-acquired pneumonia
2. Inpatients from 2017 to 2019
3. Regardless of age and gender

Exclusion Criteria:

1. Patients diagnosed with hospital-acquired pneumonia
2. Patients who take two or more oral mucolytics
3. Patients with combined use of Chinese and Western expectorants other than mucolytic drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study adopts a retrospective research design to analyze the real-world data of Eucalyptol, Limonene and Pinene Enteric Soft Capsules, to evaluate the effectiveness, safety and economy of Eucalyptol, Limonene and Pinene Enteric Soft Capsules in the real clinical treatment of community-acquired pneumonia patients.
  It is estimated that approximately 10,000 subjects from the six hospitals will meet the enrollment criteria to enter this retrospective real-world study.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of cough-related symptoms improvement | 7 days
  Rate of cough-related symptoms improvement in the expectorant treatment of inpatients with community-acquired pneumonia. Compared the differences of the rates of cough improvement between the experiment group and the control group.
  The cough-related symptoms are evaluated and recorded in the inpatients' medical records. All the descriptions of cough-related symptoms and assessments in every inpatient's medical records will be captured.

SECONDARY OUTCOMES:
Rate of overal cure and improvement in pneumonia treatment | Up to 30 days
  The overal pneumonia treatment results, include cured, improved, dead and other states, are assessed and recorded in the discharge summaries. The overal cure and improvement rate calculation in every group is based on the cured and improved states.
Hospitalization length of stay | Up to 30 days
  The mean hospitalization length of stay in every group is analyzed according the discharge summaries.
Rate of pulmonary imageological improvement | Up to 30 days
  The pulmonary imageological resultes include improved, deteriorative and unchanged states. The improvement rate calculation in every group is based on the improved state according to the last imageological reports before discharge.
Rate of normalization of vital signs | 7 days
  The vital signs, include temperature, pulse and respirations, are measured during the pre and post treatment. The normalization rate of vital signs is analyzed among the patients with abnormal vital signs measurements before treatment.
Rate of normalization of inflammatory index of pneumonia | 7 days
  The Inflammatory indexes of pneumonia, include CRP, PCT, SAA, WBC, IL-6 and lymphocyte count, are measured during the pre and post treatment. The normalization rates of inflammatory indexes of pneumonia are analyzed among the patients with abnormal indexes measurements before treatment
Safety assessment: adverse events | Up to 30 days after first dose
  Assess safety through monitoring of adverse events, and the collection of conventional laboratory data. All the adverse events during the pre and post treatment will be captured.
Cost-effectiveness ratio | Up to 30 days
  The all-cause healthcare will be determined by all the costs happened during the whole hospital stays (i.e.,skilled nursing facility, total medical, prescriptions). Effectiveness will be measured by the primary outcome, the rate of cough-related symptoms improvement within 7 days. The cost-effectiveness ratio is determined by the ratio of the all-cause healthcare to the rate of cough-related symptoms improvement within 7 days.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Background] Koo HJ, Lim S, Choe J, Choi SH, Sung H, Do KH. Radiographic and CT Features of Viral Pneumonia. Radiographics. 2018 May-Jun;38(3):719-739. doi: 10.1148/rg.2018170048. PMID 29757717
- [Background] Pan F, Ye T, Sun P, Gui S, Liang B, Li L, Zheng D, Wang J, Hesketh RL, Yang L, Zheng C. Time Course of Lung Changes at Chest CT during Recovery from Coronavirus Disease 2019 (COVID-19). Radiology. 2020 Jun;295(3):715-721. doi: 10.1148/radiol.2020200370. Epub 2020 Feb 13. PMID 32053470
- [Background] Wang C, Shi QP, Ding F, Jiang XD, Tang W, Yu ML, Cheng JQ. Reevaluation of the post-marketing safety of Xuebijing injection based on real-world and evidence-based evaluations. Biomed Pharmacother. 2019 Jan;109:1523-1531. doi: 10.1016/j.biopha.2018.10.190. Epub 2018 Nov 14. PMID 30551404
- [Background] Naranjo CA, Busto U, Sellers EM, Sandor P, Ruiz I, Roberts EA, Janecek E, Domecq C, Greenblatt DJ. A method for estimating the probability of adverse drug reactions. Clin Pharmacol Ther. 1981 Aug;30(2):239-45. doi: 10.1038/clpt.1981.154. No abstract available. PMID 7249508
- [Background] Agbabiaka TB, Savovic J, Ernst E. Methods for causality assessment of adverse drug reactions: a systematic review. Drug Saf. 2008;31(1):21-37. doi: 10.2165/00002018-200831010-00003. PMID 18095744
- [Background] Fine MJ, Auble TE, Yealy DM, Hanusa BH, Weissfeld LA, Singer DE, Coley CM, Marrie TJ, Kapoor WN. A prediction rule to identify low-risk patients with community-acquired pneumonia. N Engl J Med. 1997 Jan 23;336(4):243-50. doi: 10.1056/NEJM199701233360402. PMID 8995086
- [Background] van Rensburg DJ, Perng RP, Mitha IH, Bester AJ, Kasumba J, Wu RG, Ho ML, Chang LW, Chung DT, Chang YT, King CH, Hsu MC. Efficacy and safety of nemonoxacin versus levofloxacin for community-acquired pneumonia. Antimicrob Agents Chemother. 2010 Oct;54(10):4098-106. doi: 10.1128/AAC.00295-10. Epub 2010 Jul 26. PMID 20660689
- See also: Related Info — https://kns.cnki.net/kcms/detail/detail.aspx?dbcode=CJFD&dbname=CJFDZHYX&filename=ZHJH201604008&v=qCuiG%25mmd2F6QNYtzfsAcmKWVee6oAWq7A%25mmd2F32bE%25mmd2FeyB4Sz843vxcLKscnAXXNuoEjHP38
- See also: Related Info — https://kns.cnki.net/kcms/detail/detail.aspx?dbcode=CJFD&dbname=CJFD2013&filename=HAIX201305046&v=9Bc6MSciMFxPiuSHHUHgKHy%25mmd2BB6g9VdyRglS96XjiAVg4Z3R6D%25mmd2BV%25mmd2BagbXJXq7BQmB
- See also: Related Info — https://kns.cnki.net/kcms/detail/detail.aspx?dbcode=CJFD&dbname=CJFD2011&filename=QQHB201105043&v=1Gp4My%25mmd2FD4duhXu2aD9QZl7%25mmd2BzB6fkakB16oSdSHnf54lz%25mmd2FLhI9clExLJsVkqLE6xh
- See also: Related Info — https://kns.cnki.net/kcms/detail/detail.aspx?dbcode=CJFD&dbname=CJFDLAST2015&filename=XDJH201501031&v=%25mmd2BG%25mmd2F4hJcGfPCcVOIDUUrO0hSzjW8XkEPNvnSYnjvPm3e9bJJf%25mmd2FK4ZR9KMlF3ImMEn
- See also: Related Info — https://kns.cnki.net/kcms/detail/detail.aspx?dbcode=CJFD&dbname=CJFDLAST2019&filename=ZGUD201906015&v=yFr2CoeGjL0Lk26b2lZ%25mmd2FrHIuQmQuK1qiX1440YHCv%25mmd2BmpZAy3bK%25mmd2B26WjZ9u8LBq0S
- See also: Related Info — https://kns.cnki.net/kcms/detail/detail.aspx?dbcode=CJFD&dbname=CJFDLAST2018&filename=GWZW201804019&v=ULRpRwDBDzFsFtLHuMrsxZvSAfj1bLKb%25mmd2BKzXulrceZt1%25mmd2F%25mmd2BZFNBaAA%25mmd2F4Ad9ZnhlEZ
- See also: Related Info — http://www.bjjiuhe.com/product/